CLINICAL TRIAL: NCT06931925
Title: Recall of a Cohort of Subjects in the Mediterranean Area. Monitoring of Liver Diseases (NUTRIHEP 3).
Acronym: Nutrihep3
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Dr. Rossella Donghia, Principal Investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: Nutrihep3
Record Dates: First submitted 2025-04-04; First posted 2025-04-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cohort Study
Keywords: Cohort Study; GWAS; MASLD; Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum Plasma Stool Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver diseases represent a significant public health problem, with a high prevalence and a growing incidence worldwide, and a significant impact on global morbidity and mortality, causing approximately 2 million deaths annually.

Deaths are largely attributable to complications of cirrhosis and hepatocellular carcinoma.

The most common causes of cirrhosis worldwide are related to viral hepatitis, alcohol, and non-alcoholic fatty liver disease caused by poor dietary habits.

Regarding the hepatitis B virus (HBV), the vaccination program, together with the improvement of socioeconomic conditions and greater public awareness, have progressively reduced the incidence and prevalence of this viral disease. Chronic hepatitis related to the hepatitis C virus (HCV), after an increase in the 1980s and 1990s, is showing a decreasing trend, particularly among younger age groups. While other studies have focused on liver diseases of metabolic origin, the most recent epidemiological data concerning the Italian population were collected in the late 1990s. Since a decade has now passed, it was thought that it might be interesting to collect new data on the prevalence pattern of liver diseases, especially in southern Italy, particularly in a municipality equally geographically distant from both the coast and the inland. Therefore, this observational study aims to analyze the evolution of liver diseases through the recall of a cohort of patients already identified in the Mediterranean area. The cohort is composed of individuals residing in the municipality of Putignano (BA) who have already undergone evaluation of liver function, comorbidities and dietary habits, in addition to adding genetic information through genome-wide association (GWAS) analyses, useful for identifying associations between genetic variants and specific phenotypic characteristics

DETAILED DESCRIPTION:
Liver diseases represent a significant public health problem, with a high prevalence and a growing incidence worldwide, and a significant impact on global morbidity and mortality, causing approximately 2 million deaths annually. Deaths are largely attributable to complications of cirrhosis and hepatocellular carcinoma. The most common causes of cirrhosis worldwide are related to viral hepatitis, alcohol, and non-alcoholic fatty liver disease caused by poor dietary habits. Hepatotropic viruses are the etiological factor in most cases of acute hepatitis, but drug-induced liver injury increasingly represents a significant percentage of cases.

In Italy, the incidence of liver diseases has been the subject of studies in recent years. Based on these data, Italy has been identified as a "hyper-endemic" region where both viral and metabolic etiologies are responsible for a high prevalence and incidence of chronic liver diseases. Furthermore, a progressive increase in the incidence of viral hepatitis from Northern to Southern Italy has been observed. In recent decades, the etiology of these diseases has been undergoing a significant change.

Regarding the hepatitis B virus (HBV), the vaccination program, along with improved socioeconomic conditions and greater population awareness, have progressively reduced the incidence and prevalence of this viral disease. Chronic hepatitis related to the hepatitis C virus (HCV), after an increase in the 1980s and 1990s, is now showing a decreasing trend, particularly among younger age groups. While other studies have focused on liver diseases of metabolic origin (ASLD, MetALD, ALD, etc.), which are indicated as one of the most common causes of liver disease worldwide and in Italy, the most recent epidemiological data concerning the Italian population were collected in the late 1990s. As a decade has now passed, it was thought that it might be interesting to collect new data on the prevalence pattern of liver diseases, especially in Southern Italy, particularly in a municipality geographically equidistant from both the coast and the hinterland.

Therefore, this observational study aims to analyze the evolution of liver diseases by recalling a cohort of patients already identified in the Mediterranean area. The cohort consists of individuals residing in the municipality of Putignano (BA) who have already undergone evaluation of liver function, comorbidities, and dietary habits, in addition to adding genetic information through genome-wide association (GWAS) analysis, useful for identifying associations between genetic variants and specific phenotypic characteristics with the aim of discovering genetic correlations that can contribute to the molecular understanding of liver diseases and related comorbidities, using a representative population sample.

The analysis of the collected data aims to identify risk factors and predictive biomarkers of liver disease progression, with the goal of optimizing prevention and management strategies. The results will provide useful information to improve clinical surveillance and promote personalized interventions in individuals with liver diseases. The analyses will be conducted using advanced bioinformatics and statistical methodologies to ensure the robustness of the results.

This recall will be carried out almost 20 years after the first one. The recall of subjects will allow for a longitudinal assessment of disease progression factors or the onset of the disease.

The aim of this cohort study is not only to recall subjects previously involved in the Nutrihep 1 and Nutrihep2 Studies, but, like all cohort studies, to evaluate the association between an exposure and an outcome in a group of individuals. Furthermore, in addition to re-evaluating the parameters previously considered (blood tests, dietary questionnaire, and physical activity) in order to study their variation, and whole-genome genotyping will performe Whole-genome genotyping of single nucleotide polymorphisms (SNPs) will be performed using high-throughput genomic technologies, such as SNP-array technology. This technology allows for the analysis of thousands/millions of genetic variants evenly distributed across the entire genome, previously characterized in different ancestral populations and present in the 1000 Genomes Project phase 3 database.

The characterization of these genetic variants (SNPs) will allow us to calculate, for each subject in our study cohort, genetic and polygenic risk scores determined by the combined influence of multiple genetic variants.

Specifically, the determination of genetic and polygenic risk scores will be carried out using data obtained from genome-wide association studies (GWAS) and using sophisticated biostatistical and mathematical algorithms to weight the allele counts on the variants associated with MAFLD pathology based on the ancestral origin of our patient cohort. In subsequent phases, the genetic and polygenic risk scores will be used to study the associations with the clinical characteristics of the ill subjects in order to identify subgroups of patients with distinctive clinical characteristics and predict the risk of onset and evolution of the pathology.

The NUTRIHEP cohort (Putignano) was first established in 2006-2007, comprising a cohort of 2300 subjects, recalled from the lists of general practitioners in the municipality of Putignano (BA) with a 1:3 step.

In 2015-2018, the same subjects were recalled, with a follow-up adherence of 65.60%. Furthermore, 102 deaths were recorded from 2007 to 2014.

The recall will consider the 2300 from the 1st wave, from which the deaths evaluated through the consultation of the Death Registers via the regional EDOTTO system and those who moved to other regions will be subtracted.

Furthermore, an embedded cohort will be created to maintain the representativeness of the study population, extracted with a 1:3 step based on the registrations of general practitioners. This approach is useful because the initial cohort has aged and therefore no longer includes individuals belonging to the younger age groups, which were present at the beginning of the study but have aged over time. This allows us to maintain the age distribution similar to the initial one, preventing the cohort from becoming progressively skewed towards older age groups, as well as reducing the bias due to the aging of the cohort itself and improving the generalizability of the results. It also allows us to preserve the statistical power of the study, because especially some older age groups are critical for the analysis of the effects of exposure on the outcome.

With similar modalities to the previous ones, this observational study will focus mainly on the following phases:

Initial phase

* Creation of a list of subjects to be called, drawing from both the names of the participants in the NUTRIHEP 1 study and the residents of the Municipality of Putignano through the list of general practitioners to compensate for the younger age group;
* Re-contacting the subjects still alive, through letters sent to their home and calls;
* Scheduling appointments.

V1:

* Signing informed consent;
* Evaluation of liver health through non-invasive examination with Fibroscan;
* Anamnesis based on epidemiological parameters (age, gender, income, pathological and family history of liver-related diseases);
* Collection of anthropometric parameters such as weight, height, waist circumference, hip circumference, neck circumference, wrist circumference, and calf circumference. Furthermore, blood pressure parameters (systolic and diastolic) and physical fitness status will be recorded through the following field tests: handgrip, Sit and Reach Test, single leg stand, 30'' sit to stand, Ruffier test, VO2 max.

Enrolled subjects will be given an accelerometer that provides objective and reliable information on physical activity (accelerations, movements...) and sleep quality. It will be given on the day of recruitment and returned after 7 days.

To better understand, before the start of the project, aspects that could interfere with the success of the proposed interventions, subjects will complete an additional questionnaire:

Furthermore, tests will be completed to evaluate sleep quality and Kinesophobia, the Pittsburgh Sleep Quality Index (PSQI) and the Tampa Scale of Kinesiophobia (TSK). For the classification of sarcopenia, the Short Physical Performance Battery (SPPB) test will be administered; - Blood sampling for routine analyses. The following will be measured on the samples: complete blood count, CRP, total proteins, ceruloplasmin, alpha 1 antitrypsin, glucose, Hemoglobin A1c (Hba1C), urea, creatinine, Estimated Glomerular Filtration Rate (eGFR), total and direct bilirubin, albumin, Aspartate Aminotransferase (AST/GOT),Alanine Aminotransferase (ALT/GPT), Gamma-Glutamyl Transferase (GGT), sodium, potassium, calcium, phosphorus, iron, cholesterol, High-Density Lipoprotein (HDL), Low-Density Lipoprotein (LDL), triglycerides, cortisol, c-peptide, vitamin D, insulin, ferritin, folate, vitamin B12, parathyroid hormone, Thyroid-Stimulating Hormone (TSH), Free Triiodothyronine (FT3), Free Thyroxine (FT4), Insulin-like Growth Factor 1 (IGF-1), high-sensitivity C-reactive protein (hsCRP), pro-B-type Natriuretic Peptide (proBNP), zinc, magnesium, HBV and HCV; Serum aliquots, possibly remaining after the routine blood chemistry analyses, will be stored in the Biobank for subsequent analyses and possibly, with the subject's consent, used for other studies that the IRCCS "Saverio de Bellis" will activate.

Genotyping analyses will be carried out on whole blood aliquots, also possibly remaining after routine analyses. Anonymity will be guaranteed by assigning a unique code to the patient at the time of enrollment.

- Delivery of self-completion questionnaires: food questionnaire (EPIC), physical activity (IPAQ, long form) and questionnaires to assess psychological health: PSS-10 (Perceived Stress Scale), H.A.D.S. (Hospital Anxiety and Depression Scale), TMI-I (Test your Memory).

V2 (7 days later):

* Collection of blood chemistry tests;
* Delivery of stool and urine samples. Fecal calprotectin and occult blood will be measured on the stool samples; Stool and urine samples will subsequently be stored in the biobank. Stool samples will be used for the evaluation of the intestinal microbiota and fecal metabolome. Urine samples will be used for metabolomics measurements; For the evaluation of the intestinal microbiota, total bacterial metagenomic DNA will be extracted from stool samples using the QIAamp FAST DNA Stool Mini Kit (Qiagen, Hilden, Germany). Microbiome characterization will be carried out using a DNA metabarcoding and shotgun metatranscriptomics approach. DNA metabarcoding analysis will be conducted using the V5-V6 hypervariable regions of 16S rRNA for bacteria (MiSeq-Illumina platform). Samples that are significant in the DNA metabarcoding analysis will be subjected to metatranscriptomics analysis (NextSeq 500 - Illumina platform). Metagenomics and metatranscriptomics data will be analyzed using bioinformatics pipelines.

To perform metabolomics tests, samples will be analyzed for volatile organic compounds (VOCs) which will be thermally desorbed by immediately transferring the fiber into the heated injection port (220 °C) of a Clarus 680 (Perkin Elmer, Beaconsfield UK) equipped with an Rtx-WAX column (30 m × 0.25 mm i.d., 0.25 µm film thickness) (Restek) and coupled to a Clarus SQ8MS (Perkin Elmer) with source and transfer line temperatures maintained at 250 and 210 °C, respectively.

* Collection of the accelerometer;
* Delivery of questionnaires and discussion of them to avoid misunderstandings and missing data.

ELIGIBILITY:
Inclusion Criteria:

* >18 Years
* Resident of Putignano (BA -Italy)

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The NUTRIHEP cohort (Putignano) was first established in 2006-2007, comprising a cohort of 2300 subjects, recalled from the lists of general practitioners in the municipality of Putignano (BA) with a 1:3 step.
  In 2015-2018, the same subjects were recalled, with a follow-up adherence of 65.60%. Furthermore, 102 deaths were recorded from 2007 to 2014.
  The recall will consider the 2300 from the 1st wave, from which the deaths evaluated through the consultation of the Death Registers via the regional EDOTTO system and those who moved to other regions will be subtracted.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Elaboration of Poligenic Risk | 36 months
  Identification of SNP groups associated with liver disease to construct a polygenic risk score

CONTACTS AND LOCATIONS:
Overall Officials: Rossella Donghia, Biologyst, Principal Investigator — IRCCS "Saverio de Bellis" - Castellana Grotte (BA) - Italy

IPD SHARING:
Plan to Share IPD: Yes
Publications on international journal

REFERENCES:
- [Background] Devarbhavi H, Asrani SK, Arab JP, Nartey YA, Pose E, Kamath PS. Global burden of liver disease: 2023 update. J Hepatol. 2023 Aug;79(2):516-537. doi: 10.1016/j.jhep.2023.03.017. Epub 2023 Mar 27. PMID 36990226
- [Background] Stroffolini T. The changing pattern of hepatitis B virus infection over the past three decades in Italy. Dig Liver Dis. 2005 Aug;37(8):622-7. doi: 10.1016/j.dld.2005.02.010. PMID 15996630
- [Background] Bedogni G, Miglioli L, Masutti F, Tiribelli C, Marchesini G, Bellentani S. Prevalence of and risk factors for nonalcoholic fatty liver disease: the Dionysos nutrition and liver study. Hepatology. 2005 Jul;42(1):44-52. doi: 10.1002/hep.20734. PMID 15895401